CLINICAL TRIAL: NCT01109446
Title: Treatment of Lateral Epicondylitis. Platelet Rich Plasma vs. Steroid vs. Saline Solution
Brief Title: Treatment of Lateral Epicondylitis: Platelet Rich Plasma Versus Steroid Versus Saline Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP RCT
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis; Tennis Elbow; Epicondylitis Lateralis
MeSH Terms: conditions — Tennis Elbow | interventions — Platelet Count; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Platelet Rich Plasma (Experimental)
  Interventions: Biological: Platelet Rich Plasma
- Isotonoic Saline Solution (Sham Comparator)
  Interventions: Procedure: Isotonic Saline Solutions
- Steroid (Triamcinolonacetonid) (Active Comparator)
  Interventions: Drug: Triamcinolonacetonid

INTERVENTIONS:
Biological: Platelet Rich Plasma — 27ml of autologous whole blood added to 3ml of ACD-A (Citrate Anticoagulant). After separation of the platelets, a high concentration of platelets (3-4ml Platelet Rich Plasma) is injected into the tendon through 7 perforations of the tendon, guided by ultrasound.
  Other Names: Plasma, Platelet Rich; PRP; Blood Platelets
  Arms: Platelet Rich Plasma
Procedure: Isotonic Saline Solutions — 3ml of Isotonic Saline Solution is injected into the tendon through 7 perforations of the tendon, guided by ultrasound.
  Other Names: Physiological Saline Solution
  Arms: Isotonoic Saline Solution
Drug: Triamcinolonacetonid — Triamcinolonacetonid 40mg/ml. 40mg of Triamcinolonacetonid is mixed with 2ml of Lidocaine 10mg/ml. It is injected deep into the tendon, guided by ultrasound.
  Other Names: Kenalog
  Arms: Steroid (Triamcinolonacetonid)

SUMMARY:
We wish to address the efficacy and safety of Platelet Rich Plasma (blood platelets), a new treatment for lateral epicondylitis (tennis elbow) and compare this new treatment to either injection with steroid or saline solution.

All injections are guided by ultrasonography.

DETAILED DESCRIPTION:
Plate Rich Plasma (PRP) is a new treatment for tendinopathy. A high concentration of blood platelets is made from the patients own blod, and then injected into the tendon. The idea is that the complex mixture of growth factors within the platelets can stimulate the healing process of the tendon. We want to address the efficacy and safety of this new treatment and compare it to either the best documented treatment, Steroid injection, or to a saline solution. We want to make a randomized controlled trial with 60 participants, 20 in each of the 3 groups, and a 12 months follow up. All injections are guided by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Duration of tennis elbow > 6 months
* Doppler activity on ultrasonography
* Lateral elbow pain that is maximal over the lateral epicondyle, and increases with pressure on the lateral epicondyle, and resisted dorsiflexion and/or middle finger.

Exclusion Criteria:

* Inflammatory disease.
* Fibromyalgia.
* Pain in hand or shoulder/neck in the same arm as being treated.
* Anticoagulation treatment.
* Wounds around the elbow.
* Treatment with steroids within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Changes in pain as a continuous outcome measure. Using The Patient-Rated Tennis Elbow Evaluation (PRTEE) questionaire. | first day, 1 months, 3 months, 6 months, 12 months.
  We use the PRTEE questionaire, which is validated for tennis elbow.

SECONDARY OUTCOMES:
Functional Disability | First day, 1 month, 3 months, 6 months, 12 months
  We use the PRTEE questionaire, validated for tennis elbow.
Ultrasonographic changes | first day, 1 months, 3 months, 6 months, 12 months
  We meassure ultrasonographic changes in: tendon thickness and doppler activity.
Adverse events | through out the entire 12 months
  The number of adverse events leading to withdrawal
Pain induced by the treatment | 1 months after treatment
  A numeric scale 0-10 adressing if the treatment caused any aditional pain, and the duration: <1 week, 1-2 week, 3-4 weeks, > 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Silkeborg Regional Hospital Department of Reumatology, Silkeborg, Denmark